CLINICAL TRIAL: NCT04671524
Title: Investigation of the Effect of Improvement in Function on Foot Pressure, Balance and Gait in Children With Rheumatic Diseases Whose Upper Extremity Affected
Brief Title: The Effect of Improvement in Function on Foot Pressure, Balance and Gait in Children With Upper Extremity Affected
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Gokce Leblebici, Physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IstanbulUC_34_2
Record Dates: First submitted 2020-12-05; First posted 2020-12-17 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-04

CONDITIONS: Upper Extremity Dysfunction; Gait, Unsteady; Juvenile Idiopathic Arthritis; Balance
Keywords: Upper Extremity; Physiotherapy; Exercise; Gait; Balance
MeSH Terms: conditions — Gait Disorders, Neurologic; Arthritis, Juvenile; Motor Activity

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- pediatric patients diagnosed with rheumatic diseases. (Experimental): Exercise group; a combination of stretching, range of motion, and strengthening exercise.
  The exercise program will take 8 weeks, 3 days per week, and 45 minutes.
  Interventions: Other: Exercise protocol
- healthy controls (No Intervention): The healthy control group will be examined and the outcomes will be compared with the experimental group.

INTERVENTIONS:
Other: Exercise protocol — a combination of stretching, range of motion, and strengthening exercise.
  Arms: pediatric patients diagnosed with rheumatic diseases.

SUMMARY:
It has been shown that movements of the upper extremity during walking are associated with lower extremity mobility. For example, when walking at a slow pace, the swing frequency of the arms is 2: 1 compared to the legs, while the limb frequency decreases to 1: 1 as the walking speed increases. That is, in order to walk fast, the lower extremity takes advantage of the acceleration of the upper extremity [1]. It is known that the muscles of the shoulder girdle also support this oscillating movement in the upper extremity during walking. Thus, it is thought that blocking or restricting shoulder girdle and arm movements during walking increases energy expenditure and heart rate, decreases gait stability, and decreases stride length and walking speed [2,3]. However, the possible effects that the upper limb can aid in movement include decreasing vertical displacement of the center of mass, decreasing angular momentum or decreasing ground reaction moment, and increasing walking stability [2-4]. In these studies that restrict arm swing, methods such as crossing the arms on the chest [5], holding the arm in a sling or pocket [6], or fixing the arms to the trunk with a bandage [7] were used. Studies have generally been conducted on healthy individuals or on the biomechanical model, and arm swing during walking has not been investigated in pathologies with only upper extremity involvement (upper extremity fractures, Juvenile Idiopathic Arthritis) without any problems with lower extremity and/or walking.

This study is aimed to reveal the effects of decreased upper extremity functionality on walking and balance.

DETAILED DESCRIPTION:
It has been shown that movements of the upper extremity during walking are associated with lower extremity mobility. For example, when walking at a slow pace, the swing frequency of the arms is 2: 1 compared to the legs, while the limb frequency decreases to 1: 1 as the walking speed increases. That is, in order to walk fast, the lower extremity takes advantage of the acceleration of the upper extremity [1]. It is known that the muscles of the shoulder girdle also support this oscillating movement in the upper extremity during walking. Thus, it is thought that blocking or restricting shoulder girdle and arm movements during walking increases energy expenditure and heart rate, decreases gait stability, and decreases stride length and walking speed [2,3]. However, the possible effects that the upper limb can aid in the movement include decreasing vertical displacement of the center of mass, decreasing angular momentum or decreasing ground reaction moment, and increasing walking stability [2-4]. In these studies that restrict arm swing, methods such as crossing the arms on the chest [5], holding the arm in a sling or pocket [6], or fixing the arms to the trunk with a bandage [7] were used. Studies have generally been conducted on healthy individuals or on the biomechanical model, and arm swing during walking has not been investigated in pathologies with only upper extremity involvement (upper extremity fractures, Juvenile Idiopathic Arthritis) without any problems with lower extremity and/or walking.

Studies performed in pathologies where upper extremity mobility and arm swing are affected have shown that the kinetic and kinematic parameters of walking are also affected [8-11]. This change in walking dynamics also changes foot pressure behavior. In a study investigating the effect of arm swing on the affected side on walking in hemiplegic individuals, ground reaction forces on the affected and unaffected sides by foot pressure analysis were examined and it was found that the maximum forces applied during the first contact and toe-off on both sides decreased [12]. In addition, the stance phase duration was higher in hemiplegic patients compared to healthy controls in both lower extremities [12]. This suggests that the affected upper extremity may change the time to transfer weight while walking. In a study investigating the changes in gait parameters in patients with brachial plexus [13] in which ground reaction forces were examined, different gait phase durations and maximum ground reaction force times were found in the affected lower extremity compared to the unaffected side. In a study examining whether the degree of upper extremity functionality has an effect on walking in patients with hemiparetic cerebral palsy; Patients were included in the exercise program aimed at increasing upper extremity function, and as a result, it was found that while upper extremity function increased, patients improved walking parameters and walking distance [14]. Zhou et al. investigated the effects of an active upper extremity exercise program in patients with spinal cord injuries and demonstrated the usefulness of active upper extremity participation in walking [15].

With these results in the literature, the effect of reduced upper extremity function on gait and balance in disease groups (such as rheumatic diseases with only upper extremity involvement, upper extremity fractures) without affecting walking or any neurological/orthopedic diagnosis that may affect walking was not investigated.

The aim of this study is to reveal the effects of decreased upper extremity functionality on walking and balance.

ELIGIBILITY:
Inclusion Criteria:

* To be in the 10-18 ages group (In order for the devices to comply with the minimum measurement criteria and to be able to cooperate with the study)
* Being diagnosed with rheumatic diseases at least 6 months ago with only upper extremity affected
* Unilateral upper extremity involvement

Exclusion Criteria:

* Having an acute pathology that could affect walking
* To be diagnosed with orthopedic/neurological pathology that will affect work and cooperation

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 39 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Fall risk | immediately after exercise protocol
  These test results will be evaluated with Biodex Balance device. The test trials are completed on the device at two different conditions, eyes open comfortable stance and eyes closed comfortable stance. The outcome is the sway variation index (SVI).
Postural Stability | immediately after exercise protocol
  These test results will be evaluated with Biodex Balance device. The test trials are completed on the device at one condition, eyes open, and automatic foot placement stance. The outcome is the stability index.
Bilateral Comparison | immediately after exercise protocol
  These test results will be evaluated with Biodex Balance device. The test trials are completed on the device at two different conditions, the right leg stance and left leg stance. The outcome is the sway index.
Single limb stance | immediately after exercise protocol
  This outcome will be evaluated with foot pressure analysis. The time between first and second peak forces during walking is the single-limb stance duration.

SECONDARY OUTCOMES:
Arm Swing Amplitude | immediately after exercise protocol
  The difference between the maximum flexion and extension of the shoulder is the arm swing amplitude during walking. The arm swing amplitude will be evaluated 2-dimensionally with the help of the Kinovea video player.
Jebsen-Taylor Hand Function Test | immediately after exercise protocol
  The Jebsen-Taylor Hand Function Test (JTHFT) is a standardized and objective measure of fine and gross motor hand function using simulated activities of daily living (ADL). The outcome is the sum of time taken for each sub-test, which is rounded to the nearest second.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University-Cerrahpaşa, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wagenaar RC, van Emmerik RE. Resonant frequencies of arms and legs identify different walking patterns. J Biomech. 2000 Jul;33(7):853-61. doi: 10.1016/s0021-9290(00)00020-8. PMID 10831760
- [Background] Bruijn SM, Meijer OG, Beek PJ, van Dieen JH. The effects of arm swing on human gait stability. J Exp Biol. 2010 Dec 1;213(Pt 23):3945-52. doi: 10.1242/jeb.045112. PMID 21075935
- [Background] Meyns P, Bruijn SM, Duysens J. The how and why of arm swing during human walking. Gait Posture. 2013 Sep;38(4):555-62. doi: 10.1016/j.gaitpost.2013.02.006. Epub 2013 Mar 13. PMID 23489950
- [Background] Collins SH, Adamczyk PG, Kuo AD. Dynamic arm swinging in human walking. Proc Biol Sci. 2009 Oct 22;276(1673):3679-88. doi: 10.1098/rspb.2009.0664. Epub 2009 Jul 29. PMID 19640879
- [Background] Pontzer H, Holloway JH 4th, Raichlen DA, Lieberman DE. Control and function of arm swing in human walking and running. J Exp Biol. 2009 Feb;212(Pt 4):523-34. doi: 10.1242/jeb.024927. PMID 19181900
- [Background] Kuhtz-Buschbeck JP, Jing B. Activity of upper limb muscles during human walking. J Electromyogr Kinesiol. 2012 Apr;22(2):199-206. doi: 10.1016/j.jelekin.2011.08.014. Epub 2011 Sep 25. PMID 21945656
- [Background] Yizhar Z, Boulos S, Inbar O, Carmeli E. The effect of restricted arm swing on energy expenditure in healthy men. Int J Rehabil Res. 2009 Jun;32(2):115-23. doi: 10.1097/MRR.0b013e32830d3675. PMID 19065107
- [Background] Behrman AL, Harkema SJ. Locomotor training after human spinal cord injury: a series of case studies. Phys Ther. 2000 Jul;80(7):688-700. PMID 10869131
- [Background] Meyns P, Van Gestel L, Massaad F, Desloovere K, Molenaers G, Duysens J. Arm swing during walking at different speeds in children with Cerebral Palsy and typically developing children. Res Dev Disabil. 2011 Sep-Oct;32(5):1957-64. doi: 10.1016/j.ridd.2011.03.029. Epub 2011 May 4. PMID 21531534
- [Background] Stephenson JL, Lamontagne A, De Serres SJ. The coordination of upper and lower limb movements during gait in healthy and stroke individuals. Gait Posture. 2009 Jan;29(1):11-6. doi: 10.1016/j.gaitpost.2008.05.013. Epub 2008 Jul 11. PMID 18620861
- [Background] Ford MP, Wagenaar RC, Newell KM. Arm constraint and walking in healthy adults. Gait Posture. 2007 Jun;26(1):135-41. doi: 10.1016/j.gaitpost.2006.08.008. Epub 2006 Sep 25. PMID 16997561
- [Background] Kim HD, Kim JG, Jeon DM, Shin MH, Han N, Eom MJ, Jo GY. Analysis of Vertical Ground Reaction Force Variables Using Foot Scans in Hemiplegic Patients. Ann Rehabil Med. 2015 Jun;39(3):409-15. doi: 10.5535/arm.2015.39.3.409. Epub 2015 Jun 30. PMID 26161347
- [Background] Grodner MR, Dudzinski K, Zdrajkowski Z, Molik A, Nosarzewska A. Selected gait parameters in children with obstetric brachial plexus injury (OBPI) - a pilot study. Ortop Traumatol Rehabil. 2012 Nov-Dec;14(6):555-68. doi: 10.5604/15093492.1024721. PMID 23382283
- [Background] Cohen-Holzer M, Sorek G, Schless S, Kerem J, Katz-Leurer M. The Influence of a Constraint and Bimanual Training Program Using a Variety of Modalities, on Upper Extremity Functions and Gait Parameters Among Children with Hemiparetic Cerebral Palsy: A Case Series. Phys Occup Ther Pediatr. 2016;36(1):17-27. doi: 10.3109/01942638.2014.990549. Epub 2014 Dec 18. PMID 25521486
- [Background] Zhou R, Alvarado L, Ogilvie R, Chong SL, Shaw O, Mushahwar VK. Non-gait-specific intervention for the rehabilitation of walking after SCI: role of the arms. J Neurophysiol. 2018 Jun 1;119(6):2194-2211. doi: 10.1152/jn.00569.2017. Epub 2018 Jan 24. PMID 29364074